CLINICAL TRIAL: NCT06793228
Title: Nanocrystalline Megestrol Combined with Immunochemotherapy As First-Line Treatment for Cachexia in Extensive-Stage Small Cell Lung Cancer: a Patient-Centered Phase II Study
Brief Title: Nanocrystalline Megestrol + Immunochemo As 1st-Line for ES-SCLC Cachexia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qiming Wang, professor, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-542
Record Dates: First submitted 2025-01-07; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: SCLC, Extensive Stage
Keywords: ES-SCLC
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- criteria-fulfilled (CF) cohort (Experimental): Patients must meet all inclusion and exclusion criteria. Erolled patients will be randomly assigned to receive Nanocrystalline Megestrol Acetate (5ml once a day, up to 12 weeks) +Tislelizumab (200mg on day 1, once every 3 weeks) combined with chemotherapy (Carboplatin, AUC=5 on day 1+ Etoposide, 100mg/m2 on day 1 to day 3, once every 3 weeks). Megestrol will be discontinued after the completion of 4 cycles. Tislelizumab 200 mg will be used as maintenance therapy, repeated every 3 weeks until disease progression or intolerable toxicity.
  Interventions: Drug: Tislelizumab
- Criteria-fulfilled(CF) cohort (Active Comparator): Patients must meet all inclusion and exclusion criteria. Erolled patients will be randomly assigned to receive Tislelizumab (200mg on day 1, once every 3 weeks) combined with chemotherapy (Carboplatin, AUC=5 on day 1+ Etoposide, 100mg/m2 on day 1 to day 3, once every 3 weeks). After 4 cycles of treatment, Tislelizumab 200 mg will be used as maintenance therapy, repeated every 3 weeks until disease progression or intolerable toxicity.
  Interventions: Drug: Nanocrystalline Megestrol Acetate
- compassionate use (CU) cohort (Other): Patients meet the inclusion criteria and main exclusion criteria, but may not meet the secondary exclusion criteria. Erolled patients will receive Nanocrystalline Megestrol Acetate (5ml once a day, up to 12 weeks) +Tislelizumab (200mg on day 1, once every 3 weeks) combined with chemotherapy (Carboplatin, AUC=5 on day 1+ Etoposide, 100mg/m2 on day 1 to day 3, once every 3 weeks). Megestrol will be discontinued after the completion of 4 cycles. Tislelizumab 200 mg will be used as maintenance therapy, repeated every 3 weeks until disease progression or intolerable toxicity.
  Interventions: Drug: Nanocrystalline Megestrol Acetate
- prospective real-world study (RWS) cohort (Other): Observe the clinical outcomes of ES-SCLC patients with pre-cachexia/cachexia receiving physician-targeted treatment (PTOC). Patients diagnozed with ES-SCLC, complicated pre-cachexia/cachexia, and are scheduled to receive chemo-immunotherapy will be included in this cohort. Erolled patients will receive Nanocrystalline Megestrol Acetate (5ml once a day, up to 12 weeks) + PD-1/L1 inhibitors + chemotherapy (Carboplatin, AUC=5 on day 1+ Etoposide, 100mg/m2 on day 1 to day 3, once every 3 weeks). Megestrol will be discontinued after the completion of 4 cycles. PD-1/L1 inhibitors will be used as maintenance therapy, repeated every 3 weeks until disease progression or intolerable toxicity.
  Interventions: Drug: PTOC

INTERVENTIONS:
Drug: Nanocrystalline Megestrol Acetate — Nanocrystalline Megestrol Acetate + Tislelizumab+ Chemotherapy (Carboplatin + Etoposide)
  Arms: Criteria-fulfilled(CF) cohort; compassionate use (CU) cohort
Drug: Tislelizumab — Tislelizumab combined with chemotherapy (Carboplatin + Etoposide)
  Arms: criteria-fulfilled (CF) cohort
Drug: PTOC — Nanocrystalline Megestrol Acetate+PD-(L)1 inhibitors+chemotherapy
  Arms: prospective real-world study (RWS) cohort

SUMMARY:
This study hypothesizes that nanocrystalline megestrol acetate can improve the cachexia condition in patients and enhance the efficacy of immunochemotherapy regimens. It plans to enroll patients newly diagnosed with extensive-stage small-cell lung cancer (ES-SCLC) who are in the pre-cachexia or cachexia stage of the cachexia trajectory. These patients will receive first-line standard immunochemotherapy combined with nanocrystalline megestrol acetate intervention. Compared to the use of the first-line standard immunochemotherapy regimen alone, the study will monitor changes in body weight and body composition, which are nutritional status indicators relative to baseline, to assess whether these changes can translate into improved survival benefits and enhanced quality of life for patients.

The objective of this clinical study are：1.To assess the change in body weight relative to baseline in malignant patients with ES-SCLC treated with a first-line standard immunochemotherapy regimen during treatment with a simultaneous co-administration of nanocrystalline megestrol supportive intervention, compared to standard treatment. 2.To assess the impact of simultaneous co-administration of nanocrystalline megestrol supportive intervention during treatment with a first-line standard immunochemotherapy regimen, compared to standard treatment, on survival benefit and quality of life in patients with ES-SCLC malignancy. 3.To explore the improvement in inflammatory and nutritional markers and changes in lymphocyte subpopulations in patients with ES-SCLC malignant disease with simultaneous co-administration of nanocrystalline megestrol supportive intervention during treatment with a first-line standard immunochemotherapy regimen, compared to standard treatment.

DETAILED DESCRIPTION:
This study employed a Phase II adaptive umbrella trial , aiming to enrich patients with ES - SCLC in the pre - cachexia or cachexia stage and provide them with the opportunity to receive potentially effective megestrol acetate treatment. To expand the scope of patients receiving treatment and enhance the understanding of the benefit - risk profile in a broader population, we established two cohorts: the criteria - fulfilled (CF) cohort, where patients need to meet all inclusion and exclusion criteria; and the compassionate use (CU) cohort, where patients meet the inclusion criteria and major exclusion criteria but may not meet the minor exclusion criteria. Concurrently, a prospective real - world study (RWS) was initiated to observe the clinical outcomes of patients in the pre - cachexia/cachexia stage receiving physician - selected treatment (PTOC).

The CF cohort plans to enroll 200 subjects, with liver metastasis (yes vs no), cachexia stage (pre - cachexia vs cachexia), and ECOG PS (0 - 1 vs 2) as stratification factors. These subjects will be randomly assigned to 2 treatment groups at a 1:1 ratio:

1. Nano - Megestrol Group: Nanocrystalline megestrol (QD, up to 12 weeks) + tislelizumab (Q3W, 4 cycles) + chemotherapy (carboplatin + etoposide, Q3W, 4 cycles);
2. Standard Control Group: Tislelizumab (Q3W, 4 cycles) + chemotherapy (carboplatin + etoposide, Q3W, 4 cycles).

In the CU cohort, the treatment plan and visits are consistent with the nanocrystalline megestrol group in the criteria - fulfilled (CF) cohort.In the RWS cohort, immunotherapy can use PD - 1/PD - L1 inhibitors other than tislelizumab, and other drugs are consistent with the nanocrystalline megestrol group in the criteria - fulfilled (CF) cohort.

CU and RWS groups do not set a specific number of subjects to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Good compliance and voluntary signing of a written informed consent form (ICF).
2. Age at enrolment ≥18 years, ≤75 years, and gender-neutral (patients >75 years old will be enrolled in the RWS cohort).
3. Eastern Cooperative Oncology Group (ECOG) physical status score of 0-2 (patients with PS 3 and above due to oncological factors can be enrolled in the CU cohort or RWS cohort).
4. Expected survival ≥ 6 months.
5. Patients with histologically or cytologically confirmed small cell lung cancer (SCLC) and confirmed extensive stage small cell lung cancer based on AJCC 8th edition staging or the American Legion Lung Cancer Association (VALG) Stage II staging method (excluding mixed small cell lung cancer).
6. Subjects have not received prior systemic systemic chemotherapy for metastatic disease. Subjects with prior adjuvant/neoadjuvant chemotherapy or radical synchronous or sequential radiotherapy for non-metastatic disease with curative intent are eligible for this study if disease progression occurred >6 months after the end of the last treatment.
7. Have at least one measurable tumour lesion according to RECIST v1.1.
8. Meet the diagnostic criteria for premalignant or malignant stage. Diagnostic criteria for pre-Cachexia stage

   Referring to the 2016 ESPEN consensus on terminology, the following conditions are also met:
   * Maximum weight loss <5% relative to baseline 6 months ago;

     * Anorexia (presence of anorexia complaints or anorexia/malignant condition subscale FAACT-A/CS score ≤37); (iii) Serum C-reactive protein CRP ≥ 5 mg/L. Diagnostic criteria for cachexia Any one of the following conditions combined with loss of appetite or systemic inflammatory response.

   Involuntary weight loss >5% in the last 6 months. ② Weight loss >2% when BMI <18.5kg ③ Weight loss >2% with muscle loss.
9. Determine good organ function by the following requirements:

   a) Routine haematology (no supportive therapy with any blood components and cell growth factors within 7 days prior to initiation of study treatment): i. Absolute neutrophil ANC ≥ 1.5 × 10^9/L (1,500/mm3); ii. Platelet count ≥ 100 × 10^9/L (100,000/mm3); and iii. Haemoglobin ≥ 90 g/L.

   b) Renal function: i. Creatinine clearance* (CrCl) calculated ≥ 50 mL/min

   * The Cockcroft-Gault formula will be used to calculate CrCl (Cockcroft-Gault formula) CrCl (mL/min) = (140 - age) × weight (kg) × F}/ (SCr (mg/dL) × 72) F = 1 for males; F = 0.85 for females; SCr = serum creatinine. ii. urine protein ≤ 1+ or 24-hour (h) urine protein quantitatively < 1.0 g. c) Liver function: i. serum total bilirubin (TBil) ≤ 1.5 × upper limit of normal (ULN); TBil ≤ 3 × ULN for patients with liver metastases or evidence of confirmed/suspected Gilbert's disease.

   ii. AST and ALT ≤ 2.5 × ULN; for patients with liver metastases, AST and ALT ≤ 5 × ULN iii. serum albumin (ALB) ≥ 28 g/L d) Coagulation: International Normalised Ratio and Activated Partial Thromboplastin Time ≤ 1.5 × ULN (unless the patient is on anticoagulant therapy and the coagulation parameters (PT/INR and APTT) are in the expected range for treatment with anticoagulants at screening).

   e) Cardiac function: left ventricular ejection fraction (LVEF) ≥50%.
10. Lung function indices 1st second forced expiratory volume (FEV1) >1L or >30% of predicted value, and lung carbon monoxide diffusion function (DLCO) >30% of predicted value;
11. Female patients of childbearing potential must have a urine or serum pregnancy test (if the urine pregnancy test result is not confirmed negative, a serum pregnancy test is required, and the serum pregnancy result will be used as the basis for the negative result) performed within 3 days prior to the first dose of the drug, and the result is negative. If a female patient of childbearing potential engages in sexual intercourse with an unsterilised male partner, the patient must be using an acceptable method of contraception from the start of screening and must agree to continue to use the adopted method of contraception for a period of 120 days after the last dose of study drug; the decision on whether or not to discontinue contraception after this time point should be discussed with the investigator. If an unsterilised male patient has sexual intercourse with a female partner of childbearing potential, the patient must use an effective method of contraception from the start of screening until the 120th day after the last dose of study medication; discontinuation of contraception after this time point should be discussed with the investigator.
12. The patient is willing and able to comply with the schedule of visits, treatment regimens, laboratory tests, and other requirements of the study.

Exclusion Criteria:

Subjects meeting any of the exclusion criteria baseline will be excluded from the study:

Main exclusion criteria

1. Presence of malignant conditions other than those caused by oncological etiology such as chronic respiratory failure requiring home oxygen support, chronic obstructive pulmonary disease, chronic and persistent congestive heart failure, acquired immunodeficiency syndrome, uncontrollable thyroid disease.
2. Presence of any condition that interferes with gastrointestinal absorption such as dysphagia, malabsorption, previous history of gastrectomy, or uncontrollable vomiting; being on tube feeding or parenteral nutrition; presence of anorexia nervosa, anorexia due to psychiatric disorders, or pain that makes it difficult to eat.
3. Being on other appetite or weight-increasing medications such as: adrenocortical steroids (except for short-term use of dexamethasone during chemotherapy), androgens, progesterone analogues, thalidomide, and anamorelin or other appetite stimulants.
4. Use of any proprietary or herbal medicine used for cancer control within 14 days prior to the first dose of study drug.
5. Pre-existing (within 3 years) or current other malignancies, except cured localised tumours (e.g. basal cell skin cancer, squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ, etc.).
6. Concurrent enrolment in another clinical study, unless it is an observational, non-interventional clinical study or a follow-up period of an interventional study.
7. Previous treatment with any other antibody or drug specifically targeting the T-cell co-stimulatory or checkpoint pathway such as anti-PD-1, PD-L1 or CTLA-4 therapy.
8. Presence of esophagogastric fundal varices, severe ulcers, history of gastrointestinal perforation and/or fistulae, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), history of intra-abdominal abscess or acute gastrointestinal bleeding, thromboembolic disease, ascites, or lower extremity oedema in the 6 months prior to the first dose.
9. Current uncontrolled co-morbidities including, but not limited to, decompensated cirrhosis, renal failure, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis, or psychiatric/social conditions that would limit the patient's ability to comply with the requirements of the study or affect the patient's ability to provide written informed consent.
10. Pre-existing history of myocarditis, cardiomyopathy, or malignant arrhythmia. Unstable angina requiring hospitalisation, myocardial infarction, congestive heart failure (aortic aneurysm of grade 2 and at risk of rupture as determined by the New York Heart Association functional class), or other cardiac impairment (e.g., poorly controlled arrhythmia, myocardial ischaemia) that may interfere with the evaluation of the safety of the investigational drug, within 6 months prior to the first dose of study drug.
11. Severe chronic or active infection (including tuberculosis infection, etc.) requiring systemic antibacterial, antifungal, or antiviral therapy ≤ 14 days prior to the first dose of study drug.
12. Patients with active molluscum contagiosum metastases, or brain metastases that are not well controlled; Patients with stable treated brain metastases may be enrolled at the discretion of the investigator; Patients with untreated, asymptomatic brain metastases may be enrolled at the judgement of the investigator, but will require regular brain imaging of the disease site.
13. Major surgical procedure or serious trauma within 30 days prior to the first dose of the drug or major surgical procedure planned within 30 days of the first dose of the drug.
14. Live or live attenuated vaccine administered within 30 days prior to the first dose or planned to be administered during the study period; inactivated vaccines are permitted.
15. Known hypersensitivity to any component of the study drug.
16. Females who are pregnant or breastfeeding.
17. Patients who, in the judgement of the investigator, may have poor compliance with the procedures and requirements of the study; patients who, in the judgement of the investigator, have any condition that endangers patient safety or interferes with the assessment of the study (e.g., patients treated with radiotherapy/synchrotron radiotherapy during the immunochemotherapy phase, except during the maintenance phase).

Secondary exclusion criteria (CU cohort may be included)

1. Active autoimmune disease requiring systemic therapy within the last two years, active or previous history of definite inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis or chronic diarrhoea).
2. Patients with Cushing's syndrome, adrenal or pituitary insufficiency; patients with difficult-to-control diabetes mellitus; and current hypertension with systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg treated with oral antihypertensive medications.

(3) Previous non-infectious pneumonia requiring systemic glucocorticoid therapy or current non-infectious pneumonia combined with mild to moderate interstitial pneumonia, inactive interstitial pneumonia.

4) Presence of unmitigated toxicity from prior antineoplastic therapy, with unmitigated defined as failure to recover to NCI CTCAE version 5.0 grade 0 or 1 (except alopecia areata) or failure to recover to levels specified in the inclusion/exclusion criteria.

5) History of known allogeneic organ transplantation and allogeneic haematopoietic stem cell transplantation; history of organ or haematopoietic stem cell transplantation requiring immunosuppression.

6) Patients with chronic hepatitis B or chronic hepatitis B virus carriers with HBV DNA ≥500 IU/mL (2500 copies/mL), or hepatitis C patients.

7) Other circumstances as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
The proportion of weight increase relative to baseline > 5% (Week 12) | after 12 weeks of treatment
  The proportion of weight increase relative to baseline > 5% (Week 12)

SECONDARY OUTCOMES:
Objective Response Rate | From date of randomization until the date of first documented date of death from any cause, assessed up to 60 months
  Proportion of patients with reduction in stable in tumor burden of a predefined amount，Baseline until partial response (PR) or complete response (CR), whichever occurs first，assessed up to 12 months
Progression Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time from random to either radiological progression or death
overall survival (OS ) | From date of randomization until the date of first documented date of death from any cause, assessed up to 60 months
  Time from the first treatment to death from any cause or the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Qiming Wang, Principal Investigator — Henan Cancer Hospital
Locations (4):
- China (4):
  - The First Affiliated Hospital of Henan University of Science and Technolog, Luoyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Henan cancer hospital,, Zhengzhou, Henan
  - Zhengzhou Third People's Hospital", Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No